CLINICAL TRIAL: NCT05735106
Title: Neck Circumference to Thyromental Distance Ratio As a Reliable Indicator for Predicting Difficult Intubation in Obese Patients for Elective Surgery Under General Anesthesia
Brief Title: NC/TMD Ratio As a Difficult Airway Predictor in Obese Patients
Status: Completed | Type: Observational
Sponsor: KRL Hospital, Islamabad (Other)
Responsible Party: Principal Investigator, Mahnoor Shabbir, Principle investigator, KRL Hospital, Islamabad
Other Study IDs: NC/TMD1
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Difficult / Failed Intubation
Keywords: difficult intubation; NC/TM distance ratio; intubation difficulty score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A (predicted easy intubation): Group A labelled as predicted easy intubation on the basis of NC/TM distance ratio <5
- Group B (predicted difficult intubation): Group B labelled as predicted Difficult intubation on the basis of NC/TM distance ratio ≥ 5

SUMMARY:
To assess accuracy of NC/TM distance ratio in terms of sensitivity, specificity, negative predictive value (NPV) and positive predictive value (PPV) for predicting difficult intubation in obese patient with Intubation difficulty score (IDS) as gold standard.

DETAILED DESCRIPTION:
At Preanaesthesia clinic patients , neck circumference to Thyromental distance ratios of obese patients with BMI >30Kg/m2 will be calculated and patients will be divided into two groups on the basis of Nc/TMD ratio as anticipated easy intubation ( NC/TMD<5) And anticipated difficult intubation ( NC/TMD ≥5).

Intra-operatively, patients Intubation difficulty scale score will calculated and the data obtained from IDS score will be compared with NC/TMD ratio as a predictor of difficult Intubation and diagnostic accuracy of NC/TMD as a reliable indicator of difficult intubation in obese patients will be calculated by statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I to III
2. Body Mass Index (BMI) of 30kg/m2 or more
3. age 18-65 years

Exclusion Criteria:

1. non consenting
2. ASA class greater than III,
3. patients undergoing general anesthesia without tracheal intubation or under regional anesthesia,
4. patients with upper airway pathology such as maxillofacial fractures, upper airway tumors or cervical spine fracture, obstetric patients, refusal of the patient, previous head and neck surgery or radiotherapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obese patients (BMI ≥30Kg/m2) of all genders, between age of 18 to 65 years, belonging to ASA class I-III, Undergoing elective surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-05-21 (Actual)

PRIMARY OUTCOMES:
Predictability of difficult airway | During anaesthesia induction
  At the preanaesthetic examination neck circumference to thyromental distance ratio will be caculated in obese patients with BMI ≥ 30KG/m2 and the predictability of difficult airway will be evaluated by statistical analysis

CONTACTS AND LOCATIONS:
Overall Officials: Mahnoor Shabbir, Principal Investigator — KrlH Islamabad
Locations (1):
- KRL Hospital, Islamabad, ICT, Pakistan